CLINICAL TRIAL: NCT00306176
Title: Rosiglitazone and Exercise in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: University of Athens (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1975
Record Dates: First submitted 2006-03-22; First posted 2006-03-23 (Estimated); Last update posted 2007-04-04 (Estimated); Status verified 2007-04

CONDITIONS: Type II Diabetes Mellitus
Keywords: rosiglitazone,exercise,cardiovascular risk factors
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rosiglitazone

INTERVENTIONS:
Drug: Rosiglitazone

SUMMARY:
The aim of the present study is to investigate the influence of systemic exercise, rosiglitazone administration and combined pharmaceutical and lifestyle intervention on cardiovascular risk factors

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetes mellitus
* Poor glycemic control

Exclusion Criteria:

* Heart failure
* Renal disease
* Liver disease
* Cardiovascular event

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-01; Study Completion 2006-10

PRIMARY OUTCOMES:
Cardiovascular risk factors alterations

CONTACTS AND LOCATIONS:
Overall Officials: Christos Liapis, PhD,MD, Study Chair — University of Athens,Greece
Locations (1):
- AHEPA University Hospital of Thessaloniki, Thessaloniki, Thessaloniki, Greece

REFERENCES:
- [Derived] Kadoglou NPE, Korakas E, Lampropoulos S, Maratou E, Kassimis G, Patsourakos N, Plotas P, Moutsatsou P, Lambadiari V. Plasma nesfatin-1 and DDP-4 levels in patients with coronary artery disease: Kozani study. Cardiovasc Diabetol. 2021 Aug 13;20(1):166. doi: 10.1186/s12933-021-01355-x. PMID 34389003
- [Derived] Kadoglou NP, Vrabas IS, Kapelouzou A, Angelopoulou N. The association of physical activity with novel adipokines in patients with type 2 diabetes. Eur J Intern Med. 2012 Mar;23(2):137-42. doi: 10.1016/j.ejim.2011.10.020. Epub 2011 Nov 29. PMID 22284243
- [Derived] Kadoglou NP, Vrabas IS, Sailer N, Kapelouzou A, Fotiadis G, Noussios G, Karayannacos PE, Angelopoulou N. Exercise ameliorates serum MMP-9 and TIMP-2 levels in patients with type 2 diabetes. Diabetes Metab. 2010 Apr;36(2):144-51. doi: 10.1016/j.diabet.2009.11.004. Epub 2010 Feb 9. PMID 20149706
- [Derived] Kadoglou NP, Iliadis F, Angelopoulou N, Sailer N, Fotiadis G, Voliotis K, Vitta I, Liapis CD, Alevizos M. Cardiorespiratory capacity is associated with favourable cardiovascular risk profile in patients with Type 2 diabetes. J Diabetes Complications. 2009 May-Jun;23(3):160-6. doi: 10.1016/j.jdiacomp.2007.12.008. Epub 2008 Apr 16. PMID 18413173
- [Derived] Kadoglou NP, Iliadis F, Liapis CD, Perrea D, Angelopoulou N, Alevizos M. Beneficial effects of combined treatment with rosiglitazone and exercise on cardiovascular risk factors in patients with type 2 diabetes. Diabetes Care. 2007 Sep;30(9):2242-4. doi: 10.2337/dc07-0341. Epub 2007 Jun 22. No abstract available. PMID 17586747